CLINICAL TRIAL: NCT01921491
Title: DHACM vs Other Commercially Available Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFDFU005
Record Dates: First submitted 2013-08-09; First posted 2013-08-13 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard of Care (Other): Surgical debridement of DFU, followed by collagen alginate and gauze dressing application to be changed daily by patient. Patient will practice Offloading. Reassessment weekly at office visit.
  Interventions: Device: Offloading
- Other Commercially Available Product (Active Comparator): Application of commercially available product with Dressing Application, to be changed weekly following surgical debridement. Patient will practice Offloading. If the ulcer has not closed completely, an additional application of commercially available product will be applied weekly at weeks 2-11.
  Interventions: Procedure: Dressing Application; Device: Offloading
- dHACM (Experimental): Application of dHACM with Dressing Application, to be changed weekly following surgical debridement. Patient will practice Offloading. If the ulcer has not closed completely, an additional piece of dHACM will be applied weekly at weeks 2-11.
  Interventions: Procedure: Dressing Application; Device: Offloading

INTERVENTIONS:
Procedure: Dressing Application — Application of a non-adherent dressing, a moisture retentive dressing, and a multi-layer compression dressing.
  Arms: Other Commercially Available Product; dHACM
Device: Offloading — Provision of offloading cast walker or similar sponsor-approved device. May convert into "instant total contact cast" and/or add felt/foam to supplement offloading.

SUMMARY:
The purpose of this study is to determine whether dehydrated human amnion/chorion membrane (dHACM) is more effective than another commercially available product or conservative measures alone when used to treat diabetic foot ulcers (DFUs).

DETAILED DESCRIPTION:
This is a prospective, stratified, randomized, controlled, comparative, parallel group, multi-center clinical trial comparing the proportion of ulcers completely healed by use of dehydrated human amnion/chorion membrane (dHACM) placed weekly versus placement of bioengineered skin substitute (BSS) placed weekly, versus standard of care in diabetic patients with a diabetic foot ulcer who have adequate arterial perfusion as defined in section, 2.0 (Patient Eligibility), for wound healing to the affected limb.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 or older.
2. Patient is willing to provide informed consent and is willing to participate in all procedures and follow up evaluations necessary to complete the study.
3. Patient's ulcer must be diabetic in origin and larger than 1 cm2. Note: Debridement will be done prior to randomization. Subject's informed consent for participating in this study, must be obtained prior to proceeding with sharp debridement.
4. Patients with Type 1 or Type 2 diabetes (criteria for the diagnosis of diabetes mellitus per ADA).
5. Ulcer must be present for a minimum of four weeks before enrollment/ randomization, with documented failure of conventional ulcer therapy to heal the wound. A two week run-in period will precede enrollment/ randomization in the trial to document the indolent nature of the wounds selected.
6. Additional wounds may be present but not within 3 cm of the study wound.
7. Wound must be present anatomically on the foot as defined by beginning below the malleoli of the ankle and be neuropathic in origin.
8. Patient's ulcer must exhibit no clinical signs of infection.
9. Serum Creatinine less than 3.0mg/dl within last six months.
10. HbA1c less than or equal to 12% within last 90 days.
11. Patient has adequate circulation to the affected extremity, as demonstrated by one of the following within the past 60 days:

    1. Dorsum transcutaneous oxygen test (TcPO2) with results ≥30mmHg, OR
    2. ABIs with results of ≥0.7 and ≤1.2, OR
    3. Doppler arterial waveforms, which are triphasic or biphasic at the ankle of affected leg.

Exclusion Criteria:

1. Patients presenting with an ulcer probing to tendon, muscle, capsule or bone (UT Grade IIIA-D). A positive probe-to-bone will be confirmed when bone or joint can be felt with a sterile, ophthalmological probe.
2. Patients whose index diabetic foot ulcers are greater than 25 cm2.
3. Patients considered not in reasonable metabolic control, confirmed by an HbA1c greater than 12% within previous 90 days.
4. Patients whose serum creatinine levels are 3.0mg/dl or greater within the last six months.
5. Patients with a known history of poor compliance with medical treatments.
6. Patients who have been previously randomized into this study, or are presently participating in another clinical trial.
7. Patients who are currently receiving radiation therapy or chemotherapy.
8. Patients with known or suspected local skin malignancy to the index diabetic ulcer.
9. Patients diagnosed with autoimmune connective tissues diseases.
10. Non-revascularizable surgical sites.
11. Active infection at site.
12. Any pathology that would limit the blood supply and compromise healing.
13. Patients that have received a biomedical or topical growth factor for their wound within the previous 30 days.
14. Patients who are pregnant or breast feeding.
15. Patients who are taking medications that are considered immune system modulators which could affect graft incorporation.
16. Known allergy to Gentamicin or Streptomycin, or to bovine collagen.
17. Patients with known hypersensitivity to components of any treatment used in the trial.
18. Wounds greater than one year in duration without intermittent healing.
19. Wounds improving greater than 20% over the first two weeks (run-in period) of the trial using standard of care dressing and camboot.
20. Patients taking Cox-2 inhibitors.
21. Planned use of Dakin's solution, Mafenide Acetate, Scarlet Red Dressing, Tincoban, Zinc Sulfate, Povidone Iodine solution, Mafenide Acetate, Polymyxin/Nystatin or Chlorhexidine during trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2013-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Proportion of ulcers achieving 100% epithelialization in the dHACM group vs other commercially available product and control. | 6 weeks
  Visitrak Wound Measurement System

SECONDARY OUTCOMES:
Proportion of patients achieving 100% epithelialization in dHACM group vs other commercially available product and control. | 12 weeks
  Visitrak Wound Measurement System
Cost effectiveness of each treatment modality. | 12 weeks
  Cost of product x number of visits

CONTACTS AND LOCATIONS:
Overall Officials: Charles Zelen, DPM, Principal Investigator — Professional Education and Research Institute, Inc.
Locations (2):
- United States (2):
  - St. Johns Outpatient Wound Center, Tulsa, Oklahoma
  - Professional Education and Research Institute, Inc., Roanoke, Virginia